CLINICAL TRIAL: NCT07100990
Title: A Randomized Controlled, Open-Label, Rater-Blinded Pragmatic Trial, Treatment of Inflammatory Myelitis and Optic Neuritis With Early vs Rescue Plasma Exchange (TIMELY-PLEX)
Brief Title: Treatment of Inflammatory Myelitis and Optic Neuritis With Early vs Rescue Plasma Exchange (TIMELY-PLEX)
Acronym: TIMELY-PLEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, John J Chen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-000657
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Optic Neuritis; Myelitis; Myelitis, Transverse
Keywords: Plasma Exchange; Plasmapheresis; Apheresis; Pheresis
MeSH Terms: conditions — Optic Neuritis; Myelitis; Myelitis, Transverse | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Optic Neuritis (ON) "Rescue PLEX" (Active Comparator): Adult participants presenting within 8 days of symptom onset with severe Optic Neuritis (ON) (visual acuity of 20/200 or worse
  Interventions: Drug: High-dose corticosteroids (HDCS)
- Optic Neuritis (ON) "Early PLEX" (Experimental): Adult participants presenting within 8 days of symptom onset with severe Optic Neuritis (ON) (visual acuity of 20/200 or worse
  Interventions: Drug: High-dose corticosteroids (HDCS) and PLEX
- Transverse Myelitis "Rescue PLEX" (Active Comparator): Adult participants presenting within 8 days of symptom onset with severe Transverse Myelitis (TM) (expanded Disability Status Scale [EDSS] of 3.0 or worse)
  Interventions: Drug: High-dose corticosteroids (HDCS)
- Transverse Myelitis "Early PLEX" (Experimental): Adult participants presenting within 8 days of symptom onset with severe Transverse Myelitis (TM) (expanded Disability Status Scale [EDSS] of 3.0 or worse)
  Interventions: Drug: High-dose corticosteroids (HDCS) and PLEX

INTERVENTIONS:
Drug: High-dose corticosteroids (HDCS) — Subjects will receive initial treatment with high-dose corticosteroids (HDCS) in the form of methylprednisolone (1,000mg daily) administered intravenously for 5 days or a bioequivalent dose of oral corticosteroids (e.g., 1,250mg prednisone daily or 176mg dexamethasone daily).
  Subjects will be escalated to PLEX if there is an insufficient response to HDCS (decision point at 14±2 days for the ON sub-trial and 7±2 days for the TM sub-trial) PLEX will be performed as 5 sessions over 5-10 days, with 1-1.5 plasma volumes exchanged per session.
  Other Names: Rescue Plex
  Arms: Optic Neuritis (ON) "Rescue PLEX"; Transverse Myelitis "Rescue PLEX"
Drug: High-dose corticosteroids (HDCS) and PLEX — Subjects will receive treatment with high-dose corticosteroids (HDCS) and PLEX initiated concurrently.
  HDCS will be administered in the form of methylprednisolone (1,000mg daily) administered intravenously for 5 days or a bioequivalent dose of oral corticosteroids (e.g., 1,250mg prednisone daily or 176mg dexamethasone daily).
  PLEX will be performed as 5 sessions over 5-10 days, with 1-1.5 plasma volumes exchanged per session.
  Other Names: Early Plex
  Arms: Optic Neuritis (ON) "Early PLEX"; Transverse Myelitis "Early PLEX"

SUMMARY:
The purpose of this research is to evaluate if early vs rescue Therapeutic Plasma Exchange (PLEX) treatment algorithm leads to better visual outcomes in severe Optic Neuritis and leads to better neurological disability outcomes in severe Transverse Myelitis.

ELIGIBILITY:
Study Population and Setting

The proposal will recruit participants presenting to participating sites with severe ON or severe TM to two separate sub-trials. The detailed inclusion and exclusion criteria for each sub-trial are listed below:

Optic Neuritis Sub-Trial:

Inclusion criteria:

* ≥18 years of age
* MRI orbits demonstrating evidence of new T2 hyperintensity and/or post-gadolinium contrast enhancement of the optic nerve(s) and meeting the clinical criteria for Optic Neuritis
* Visual acuity 20/200 or worse
* Within 8 days of onset of visual symptoms
* Able to initiate PLEX within 72h of the first dose of HDCS (if randomized to the "Early PLEX" treatment arm)
* Able to sign and date informed consent form
* Willingness to comply with all study procedures and availability for the duration of the study

Exclusion criteria:

* Evidence of prior episode of optic neuritis in the affected eye (by history or ophthalmological evaluation)
* Ophthalmological comorbidity that would significantly affect best corrected visual acuity or visual fields
* Pregnancy
* Presence of any contraindication to receiving HDCS or PLEX, including, but not limited to, hemodynamic instability, significant bleeding/coagulopathy, or sepsis.
* Any medical condition that, in the opinion of the investigator, may interfere with the patient's participation in the trial, pose any added risk for the patient, or confound the assessment of the patient (including but not limited to concurrent neurological disease and/or medical comorbidity)
* Treatment with any investigational agent within 6 months of baseline or five half-lives of the investigational agent (whichever is longer)
* Ongoing/prior treatment with immune-modulating/immunosuppressive therapy including:

  * Mycophenolate mofetil, azathioprine, methotrexate, fingolimod, siponimod, ponesimod, ozanimod, tocilizumab, satralizumab, eculizumab or ravulizumab within 3 months of randomization
  * Anti-CD20 (rituximab, ocrelizumab, ofatumumab, ublituximab) or anti-CD19 (inebilizumab) therapy within 6 months of randomization
  * Intravenous or subcutaneous immune globulin within 3 months of randomization
  * Plasma exchange within 3 months of randomization
  * Interferon-beta, glatiramer acetate, fumarates (dimethyl fumarate, monomethyl fumarate, diroximel fumarate) within 1 month of randomization
  * Teriflunomide use within prior 24 months
  * Systemic corticosteroid therapy (intravenous or oral; excluding inhaled or topical corticosteroids) within 1 month of randomization
  * Any previous treatment with alemtuzumab, cladribine, mitoxantrone or cyclophosphamide
* Previous treatment with any immune-modulating or immunosuppressive therapy not mentioned above within 6 months of randomization or five-half-lives (whichever is longer)

Transverse Myelitis Sub-Trial:

Inclusion criteria:

* ≥18 years of age
* Diagnosis of Transverse Myelitis (defined based on modified criteria adapted from the 2002 Transverse Myelitis Consortium Working Group; ALL are required)

  * Development of sensory, motor and/or autonomic symptomatology attributable to spinal cord dysfunction
  * Onset of symptoms to nadir >12 hours
  * Exclusion of extra-axial compressive etiology by neuroimaging
  * Demonstration of inflammation within the spinal cord by presence of intramedullary T2 lesion (post-gadolinium enhancing OR non-enhancing) on MRI
* Expanded Disability Status Scale [EDSS] ≥3.0 (excluding visual and cerebral functional systems)
* EDSS Pyramidal Functional System Score ≥ 2
* Within 8 days of onset of motor symptoms
* Able to initiate PLEX within 48h of the first dose of HDCS (if randomized to the "Early PLEX" treatment arm)
* Able to sign and date informed consent form
* Willingness to comply with all study procedures and availability for the duration of the study

Exclusion criteria:

* Pre-existing ambulatory, motor, sensory, or bowel/bladder disability of any cause that could confound trial assessments
* Fulfillment of possible, probable or definite spinal cord infarction diagnosis per proposed diagnostic criteria (Zalewski et al. JAMA Neurology 2018)
* History of radiation to the spine
* Pregnancy
* High clinical suspicion for infectious etiology of myelitis (e.g., fever, rash or other findings)
* Presence of any contraindication to receiving HDCS or PLEX, including, but not limited to, hemodynamic instability, significant bleeding/coagulopathy, or sepsis.
* Any medical condition that, in the opinion of the investigator, may interfere with the patient's participation in the trial, pose any added risk for the patient, or confound the assessment of the patient (including but not limited to concurrent neurological disease and/or medical comorbidity)
* Treatment with any investigational agent within 24 weeks of baseline or five half-lives of the investigational agent (whichever is longer)

  * Ongoing/prior treatment with immune-modulating/immunosuppressive therapy including: Mycophenolate mofetil, azathioprine, methotrexate, fingolimod, siponimod, ponesimod, ozanimod, tocilizumab, satralizumab, eculizumab or ravulizumab within 3 months of randomization
  * Anti-CD20 (rituximab, ocrelizumab, ofatumumab, ublituximab) or anti-CD19 (inebilizumab) therapy within 6 months of randomization
  * Intravenous or subcutaneous immune globulin within 3 months of randomization
  * Plasma exchange within 3 months of randomization
  * Interferon-beta, glatiramer acetate, fumarates (dimethyl fumarate, monomethyl fumarate, diroximel fumarate) within 1 month of randomization
  * Teriflunomide use within prior 24 months
  * Systemic corticosteroid therapy (intravenous or oral; excluding inhaled or topical corticosteroids) within 1 month of randomization
  * Any previous treatment with alemtuzumab, cladribine, mitoxantrone or cyclophosphamide
* Previous treatment with any immune-modulating or immunosuppressive therapy not mentioned above within 6 months of randomization or five-half-lives (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
High contrast visual acuity | 6 months
  The Optic Neuritis subjects will have high contrast visual acuity measured by ETDRS 100% high-contrast Sloan letter charts. A high contrast visual acuity of 20/20 is considered "normal," a high contrast visual acuity of 20/40 or better is required to be able to drive without restrictions, and a high contrast visual acuity of 20/200 or worse is considered legally blind.
Expanded Disability Status Score (EDSS) | 6 months
  The level of disability in Transverse Myelitis subjects will be assessed using the Expanded Disability Status Scale (EDSS). The EDSS assesses various neurological functional systems, including pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, and cereberal functions and ranges from 0 (normal neurological examination) to 10 (death). Higher scores indicate greater disability. Visual and cerebral functional system scores will be excluded from the EDSS calculation for quantification of Transverse Myelitis-related disability.

SECONDARY OUTCOMES:
Low contrast (2.5%) visual acuity | 6 months
  Optic Neuritis subjects will have low contrast visual acuity (best corrected) assessed with 2.5% low-contrast Sloan letter charts
Peri-papillary retinal nerve fiber layer (RNFL thickness) | 6 months
  Optic Neuritis subjects will have RNFL thickness measured via Retinal Optical Coherence Tomography (OCT).
Macular ganglion cell-inner plexiform layer (GCIPL) thicknesses | 6 months
  Optic Neuritis subjects will have GCIPL thickness measured via Retinal Optical Coherence Tomography (OCT).
Hardy Rand and Rittler (HRR) color plates | 6 months
  The Hardy-Rand-Rittler (HRR) color plates test will be administered to Optic Neuritis subjects. The HRR is scored based on the number of correct responses to the diagnostic plates, with the total number of correct figures out of 28 being the primary score.
National Eye Institute (NEI) 10-Item Neuro-Ophthalmic Supplement | 6 months
  Optic Neuritis subjects will complete the 10-Item Neuro-Ophthalmic Supplement, a 10-item questionnaire used to assess visual dysfunction in patients with neuro-ophthalmologic disorders. It is scored on a scale of 0 to 100, with higher scores indicating better visual functioning.
Ambulatory disability | 6 months
  Transverse Myelitis subjects will be assessed for ambulatory disability using the Hauser Ambulation Index, a timed 25 foot, 6 minute walk.
Manual dexterity (Nine-Hole Peg Test) | 6 months
  The Nine-Hole Peg Test will be administered to the Transverse Myelitis subjects. Subjects will be asked to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. They will then remove the pegs, one by one, from the board as quickly as possible. Scores are based on the time taken to complete the activity and are reported in seconds.
Patient Determined Disease Steps (PDDS) | 6 months
  Transverse Myelitis subjects will complete the Patient-Determined Disease Steps (PDDS), a self-reported disability scale with 9 levels ranging from no disability to bedridden.
Spinal Cord Injury Quality of Life questionnaire (SCI-QoL) | 6 months
  Transverse Myelitis subjects will complete the The Spinal Cord Injury Quality of Life questionnaire (SCI-QoL), which includes assessments of specific domains related to bladder/bowel dysfunction, pain, pressure ulcers, mobility/ambulation, fine motor skills, self-care, and wheelchair mobility.
PLEX Complications | 2 weeks, 1 month
  Total number of adverse events categorized according to the Common Terminology Criteria for Adverse Events v5.0
National Eye Institute (NEI) Visual Function Questionnaire (VFQ)-25 | 6 months
  Optic Neuritis subjects will complete the National Eye Institute Visual Functioning Questionnaire-25. The questionnaire consists of 25 items, covering 11 vision-related domains, plus a single global-rating item. Items are scored and converted to a 0- to 100-point scale where higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: John Chen, Principal Investigator — Mayo Clinic
Locations (25):
- United States (25):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Colorado - Anschutz Medical, Aurora, Colorado
  - Yale University School of Medicine, North Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Dean McGee Eye Institute at University of Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pittsburgh Medical Center, Magee Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials